CLINICAL TRIAL: NCT04888208
Title: Set up a Community Online in a Virtual Community Game for Tobacco Prevention in Teenagers
Brief Title: Prevention in a Virtual Community Game
Acronym: SCOTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP-INSERM
Record Dates: First submitted 2021-04-29; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-04

CONDITIONS: Tabagism
Keywords: Primary prevention; Adolescents; Internet; Empowerment; Community participation
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral (Experimental): The intervention group will benefit from discussion sessions on tobacco within the virtual world, with a group of pairs and 2 facilitators (public health researchers).
  Interventions: Behavioral: Behavioral
- Control Arm (No Intervention): The control group will be offered sources of conventional health information (government and institutional websites) on a terminal located in the virtual world.

INTERVENTIONS:
Behavioral: Behavioral — The intervention group will benefit from discussion sessions on tobacco within the virtual world, with a group of pairs and 2 facilitators (public health researchers).
  Arms: Behavioral

SUMMARY:
The main objective of the SCOTT project is to reduce tobacco experimentation of teenagers through an online intervention based on social networking and empowerment of users.

Specific objectives of this emerging project are : 1. To develop or identify an online community dedicated to teenagers where the investigators will develop anti-smoking skills and norms. It will be based on social cognitive theory and will combine multiple functionalities based on the current practices and preferences of adolescents on internet and mobile; ensuring user safety, regulatory and ethical issues ; 2. To analyse the adoption, acceptance and the usability of SCOTT among users in a limited scale 3.To develop SCOTT process and impact assessment methodology.

Research hypothesis Providing access to prevention in an online community will: 1) Strengthen anti-smoking skills 2) Enhance the empowerment of users 3) Allow the implementation of health interventions 4) Improve indicators of tobacco consumption in young people Methods The overall methodology of the project relies on a multidisciplinary approach with a consortium of French experts in public health (health promotion and epidemiology), education science, information and communication technologies, medical informatics, adolescent medicine, adolescent addictology, social sciences, ethics and law. The project will be led in 3 parts: 1) Development of the intervention - using the Integrate, Design, Assess, and Share (IDEAS) framework. Using qualitative methods (individual interview, focus groups), multidisciplinary team brainstorming, works meeting and quantitative assessment of SCOTT quality; the investigators will (a) empathize with target users, (b) specify target behavior, (c) ground in behavioral theory, (d) ideate implementation strategies, (e) prototype potential products, (f) gather user feedback, (g) build a minimum viable product, 2) Pilot study : (h) SCOTT will be deploying on a small scale to assess its usability; 3) Development of the large-scale evaluation protocol - following the recommendations of the Medical Research Council concerning the evaluation of complex interventions. The investigators will (i) develop, based on the results of the pilot test, the SCOTT process evaluation methodology, (j) develop the SCOTT impact / effectiveness evaluation methodology.

DETAILED DESCRIPTION:
Scientific context The SCOTT project stems from the "m-Health" Initiative launched in 2012 by the WHO and the International Telecommunication Union for the fight against non-communicable diseases (NCDs). The project is based on: 1) In 2014, in France, a third of high school students of all ages said they had already had the opportunity to smoke a cigarette. Smoking cigarettes is multiplied by 5 during the high school years, with one student in two who has already smoked at least once a cigarette in the last year. 2) In France the rate of computer equipment is 97% in the 12-17 and 81% have smartphones. Teenagers of 11-14 are 67% to have a social network account that they used mainly to watch videos, chat with friends and family and publish and share 3) Essential elements of risk-taking prevention programs for adolescents have been identified: using social behavior theories; using interactive skill-building methods, focusing on the social influences that encourage behavior, including peers and the media; offering multiple-component interventions; including a strong peer education or support component.

Objectives The main objective of the SCOTT project is to reduce tobacco experimentation of teenagers through an online intervention based on social networking and empowerment of users.

Specific objectives of this emerging project are : 1. To develop or identify an online community dedicated to teenagers where the investogators will develop anti-smoking skills and norms. It will be based on social cognitive theory and will combine multiple functionalities based on the current practices and preferences of adolescents on internet and mobile; ensuring user safety, regulatory and ethical issues ; 2. To analyse the adoption, acceptance and the usability of SCOTT among users in a limited scale 3.To develop SCOTT process and impact assessment methodology.

Research hypothesis Providing access to prevention in an online community will: 1) Strengthen anti-smoking skills 2) Enhance the empowerment of users 3) Allow the implementation of health interventions 4) Improve indicators of tobacco consumption in young people Methods The overall methodology of the project relies on a multidisciplinary approach with a consortium of French experts in public health (health promotion and epidemiology), education science, information and communication technologies, medical informatics, adolescent medicine, adolescent addictology, social sciences, ethics and law. The project will be led in 3 parts: 1) Development of the intervention - using the Integrate, Design, Assess, and Share (IDEAS) framework. Using qualitative methods (individual interview, focus groups), multidisciplinary team brainstorming, works meeting and quantitative assessment of SCOTT quality; the investigators will (a) empathize with target users, (b) specify target behavior, (c) ground in behavioral theory, (d) ideate implementation strategies, (e) prototype potential products, (f) gather user feedback, (g) build a minimum viable product, 2) Pilot study : (h) SCOTT will be deploying on a small scale to assess its usability; 3) Development of the large-scale evaluation protocol - following the recommendations of the Medical Research Council concerning the evaluation of complex interventions. The investigators will (i) develop, based on the results of the pilot test, the SCOTT process evaluation methodology, (j) develop the SCOTT impact / effectiveness evaluation methodology.

Expected public health impact Risk behaviors that appear in adolescence explain 17% of the total burden of disease -mainly non-communicable diseases. With SCOTT young people will gain greater control of their state of health and well-being through proactive, participatory and informative aspects of our project. Empowerment and acquisition of resilience skills will minimise the risk factors of risk behaviors, especially smoking.

Perspectives 1. To deploy and evaluate at the national level SCOTT's effectiveness in reducing experimentation and regular tobacco use among college students 2. To use data for public health research on adolescents' health and well-being in order to strengthen research towards e-health and m-health evidence using data collected from the platform and by the implementation of surveys and interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* Players of the French-speaking HABBO community;

  * Informed and consentent to the study;
  * Agreeing to complete the baseline study questionnaire.

Exclusion Criteria:

-

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
smoking behaviors perception | 4 weeks
  questionnaires build on the validated questionnaire of P2P trial (F. Coussin Gélie, BMC Public Health, 2018) derived from elements of Theory of Planned Behavior related to tabagism

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Alberti, MD, PhD, Principal Investigator — APHP
Locations (1):
- Robert Debré Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin P, Chapoton B, Bourmaud A, Dumas A, Kivits J, Eyraud C, Dubois C, Alberti C, Le Roux E. Health Promotion in Popular Web-Based Community Games Among Young People: Proposals, Recommendations, and Applications. JMIR Serious Games. 2023 Jun 9;11:e39465. doi: 10.2196/39465. PMID 37294609